CLINICAL TRIAL: NCT00466245
Title: Double-Blind, Placebo-Controlled, Dose-Finding, Phase 2 Study Assessing Safety, Tolerability, Immunogenicity of Three Dose Levels of ACAM3000 Modified Vaccinia Ankara Smallpox Vaccine in Adults With and Without Previous Smallpox Vaccination
Brief Title: Phase 2 Study of Safety, Tolerability, and Immunogenicity of Three Dose Levels of ACAM3000 Smallpox Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-249-002; NCT00170651 (obsolete NCT alias)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Smallpox
Keywords: MVA Vaccine
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A (Experimental): Previously vaccinated for smallpox, 1x10-8 dose
  Interventions: Drug: MVA Smallpox vaccine
- B (Experimental): Smallpox vaccine naive, 1x10-8 dose
  Interventions: Drug: MVA Smallpox vaccine
- C (Experimental): Previous smallpox vaccination, 1x10-7 dose
  Interventions: Drug: MVA Smallpox vaccine
- D (Experimental): Smallpox vaccine naive, 1x10-7 dose
  Interventions: Drug: MVA Smallpox vaccine
- E (Experimental): Previous smallpox vaccination, 1x10-6 dose
  Interventions: Drug: MVA Smallpox vaccine
- F (Experimental): Smallpox vaccine naive, 1x10-6 dose
  Interventions: Drug: MVA Smallpox vaccine
- G (Experimental): Previous smallpox vaccination, placebo dose
  Interventions: Drug: Placebo
- H (Experimental): Smallpox vaccine naive, placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MVA Smallpox vaccine — Two 0.5mL subcutaneous injections, separated by 28 days
  Arms: A; B; C; D; E; F
Drug: Placebo — Two 0.5mL subcutaneous injections, separated by 28 days
  Arms: G; H

SUMMARY:
A phase 2 study to assess the MVA smallpox vaccine in previously vaccinated and vaccine- naive subjects at three dose levels.

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo-controlled out-patient study conducted in multiple centers in the United States (US). Up to 700 healthy male and female adult subjects 18 to 55 years of age (inclusive), who have been previously vaccinated or subjects who are naïve to smallpox vaccine will be enrolled. Subjects will be randomized to 1 of 8 treatment groups with 100 (or 50 placebo) subjects per group in which they will receive either ACAM3000 MVA Smallpox Vaccine (1 of 3 dose levels) or placebo on Study Days 0 and 28. All personnel associated with the trial will be blinded as to treatment, with the exception of the study pharmacist who prepares the treatment for administration to each subject. There are 2 control groups in this study. A comparison of adverse events and other safety assessments between placebo and ACAM3000 MVA Smallpox Vaccine will be performed. In addition to serving as a control for safety, the previously vaccinated subjects receiving placebo will serve as a control for antibody and T-cell responses in persons with preexisting immunity who receive ACAM3000 MVA Smallpox Vaccine. Safety, tolerability, and immunogenicity data for 110 subjects undergoing primary immunization with graded doses of ACAM3000 MVA Smallpox Vaccine will be available following completion of Acambis protocol H-249-001, an ongoing phase I clinical trial. The doses levels in this study may be changed following the availability of results from protocol H-249-001. Statistical analysis will focus on comparisons among the dose levels of ACAM3000 MVA Smallpox Vaccine and comparisons of ACAM3000 MVA Smallpox Vaccine to placebo, as appropriate. A separate analysis will be performed for previously vaccinated and naïve subjects. Descriptive statistics will be used to compare demographic and baseline clinical data between stratum.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be in good general health, checked on toxicity grading table.
* for previously vaccinated subjects- must be between the ages of 33 and 55 with a previous vaccine more than 10 years ago.
* for vaccine naive subjects- must be between the ages of 18 and 32, and have never been vaccinated for smallpox.
* Female subjects must not be pregnant or lactating.

Exclusion Criteria:

* Subjects who participated in a "first responder" program.
* any history of immunodeficiency.
* any autoimmune disease
* any history of cardiac disease
* any diagnosed risk factors for ischemic coronary disease
* any history of heart palpitations or abnormalities in cardiac rhythm.
* any current or history of eczema of any description.
* Known allergy to MVA or any of its components, including eggs or egg products.
* morbid obesity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 590 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety | Study Completion

SECONDARY OUTCOMES:
Immunogenicity | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com